CLINICAL TRIAL: NCT05364229
Title: MR-guided Tumour Boost With Stereotactic Body Radiotherapy in Prostate Cancer
Brief Title: MR-guided Tumour Boost
Acronym: MRL-Boost
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-6162
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; SBRT; stereotactic body radiotherapy; tumour boost
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided Tumour Boost with SBRT (Experimental): MR-guided radiotherapy boost to MRI visible tumour
  Interventions: Radiation: MR-guided Radiotherapy Boost

INTERVENTIONS:
Radiation: MR-guided Radiotherapy Boost — IMRT/VMAT prostate whole gland SBRT to 30 Gy in 5 fractions. MRL focal boost of 15 Gy in 1 fraction will be delivered either before or after whole gland SBRT.

SUMMARY:
This is a single-arm feasibility study that is recruiting 40 patients with histologically-proven localized prostate cancer and MRI-defined lesion(s). Participants in this study will get MR-guided radiotherapy boost to MRI visible tumour before or after whole gland radiation. Participants will be followed-up as per standard of care schedule up to 5 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven localized prostate cancer.
* Low, Intermediate, and High-risk prostate cancer (ideally limited to 1 risk factor)
* Low-risk: cT1-T2a, PSA <10, and Gleason score 6
* Intermediate-risk: cT2b-c, PSA 10-20, and/or Gleason score 7
* High-risk limited to 1 risk factor: >T2, PSA >20, or Gleason score >7
* Intra-prostatic tumour(s) demonstrated on mpMRI histologically confirmed limited to =/< 1/3 total prostate volume
* Planned for EBRT (+/- ADT)
* ECOG 0 or 1
* 18 years of age or older
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Prior radiotherapy to pelvis
* Radiological evidence of regional or distant metastases at the discretion of the treating physician.
* Active ulcerative colitis or Crohn's Disease, at discretion of treating physician
* Ataxia Telangectasia and SLE
* Contraindications to MRI; including patients with pacemakers/implantable cardiac defibrillator, cerebral aneurysm clips, shrapnel injury
* Severe claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of MR-guided Linear Acceleratorfor tumour-targeted intra-prostatic dose escalation as boost | Baseline
  Total proportion of patients achieving predefined dosimetric parameters: PTV V100, PTV D90, Urethra V105, Rectum V75, Bladder V75

SECONDARY OUTCOMES:
Acute Toxicity | Baseline to 5-year follow-up
  Acute (less than or equal to 90 days) toxicity will be evaluated by using prospective follow-up and grading according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Late Toxicity | Baseline to 5-year follow-up
  Late (more than 90 days) toxicity will be evaluated by using prospective follow-up and grading according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Patient-reported quality-of-life assessed by EPIC-26 | Baseline to 5-year follow-up
  Patient-Reported Quality of Life will be assessed at baseline and at each follow-up visit (1-, 3-, and 6-months post radiation as well as years 1, 2, 3, 4, and 5) using the following assessment questionnaires: 26-Item Expanded Prostate Cancer Index Composite (EPIC-26)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada